CLINICAL TRIAL: NCT01018303
Title: Safety and Efficacy of a Novel Antioxidant-rich Multivitamin Supplement for Persons With Cystic Fibrosis
Brief Title: Safety and Efficacy of an Antioxidant-rich Multivitamin Supplement in Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Yasoo Health (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0355
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; vitamins; antioxidants; anthropometric measurements; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antioxidant-enriched multivitamin supplement (Experimental)
  Interventions: Dietary Supplement: AquADEK

INTERVENTIONS:
Dietary Supplement: AquADEK — Two AquADEK softgel vitamins on a daily basis x 12 weeks

SUMMARY:
The purpose of this study is to test the safety and efficacy of the final commercial formulation of an antioxidant enriched multivitamin supplement in softgel capsule form (AquADEKs) in increasing the plasma levels of certain nutrients and antioxidants in individuals with cystic fibrosis.

Hypothesis: An oral antioxidant-rich multivitamin supplement (AquADEKs), which uses a Generally Regarded As Safe (GRAS) molecule to form micelle-like vehicles, will safely increase systemic levels of beta-carotene, coenzyme Q10, and gamma-tocopherol, decrease PIVKA-II levels, while maintaining levels of vitamins A and D in the normal range in persons with CF > 10 years of age.

DETAILED DESCRIPTION:
In cystic fibrosis (CF), pancreatic insufficiency and a diminished bile acid pool cause malabsorption of important nutrients and dietary components leading to poor nutritional status and oxidative stress. Of particular significance is the malabsorption of fat-soluble nutrients, such as vitamins A, D, E and K which are critical for normal metabolic functions. Furthermore this malabsorption prevents individuals with CF from adequately absorbing and maintaining levels of lipophilic nutrients and antioxidants such as beta-carotene, coenzyme Q10 (CoQ10) and gamma-tocopherol which may provide benefits when supplied at levels higher than those obtained from normal diets. Current standard of care supplementation often does not normalize the blood levels of certain vitamins and antioxidants.

An oral formulation, which can form micelle-like vehicles, can be used to overcome the malabsorption of these nutrients in CF patients. A pilot study of a prototype formulation showed both safety and efficacy in increasing systemic levels of target nutrients. This study will test the safety and efficacy of the final commercial formulation (AquADEKs) in the form of a softgel capsule in increasing the plasma levels of certain nutrients and antioxidants.

Hypothesis: An oral antioxidant-rich multivitamin supplement (AquADEKs), which uses a Generally Regarded As Safe (GRAS) molecule to form micelle-like vehicles, will safely increase systemic levels of beta-carotene, coenzyme Q10, and gamma-tocopherol, decrease PIVKA-II levels, while maintaining levels of vitamins A and D in the normal range in persons with CF > 10 years of age.

Specific Aims:

1. To evaluate the safety of AquADEKs by monitoring patient reported symptoms and adverse events, and following vitamin and antioxidant levels, particularly vitamin A, to ensure that they do not exceed normative ranges after supplementation.
2. To determine the efficacy of AquADEKs in increasing the antioxidants beta-carotene, CoQ10, and γ-tocopherol and maintaining plasma levels of vitamins A, D, α-tocopherol and PIVKA-II (surrogate of vitamin K status) in the normal range.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as evidenced by a sweat chloride test > 60mEq/L or by the presence of two known CF mutations
* Male or female, ages between 10-40 years old
* > 30 kg body weight
* FEV1 > 35% predicted for age and height
* Clinically stable with no recent hospitalization within the past 2 weeks

Exclusion Criteria:

* Significant liver disease as defined by clinical findings of portal hypertension or cirrhosis or AST, ALT, or GGT >2x upper limits of normal within the previous 6 months
* Poor compliance with medical regimen as assessed by CF clinic care providers
* Oral supplementation with AquADEKs or another source of beta-carotene or CoQ10 in the 2 months prior to the study
* Pregnant or lactating
* Participation in another interventional clinical trial within the previous 2 weeks
* Difficulty swallowing softgels

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Plasma levels of beta-carotene | 12 weeks

SECONDARY OUTCOMES:
Plasma levels of coenzyme Q10, retinol (Vitamin A), 25-hydroxy vitamin D, alpha- and gamma-tocopherols (Vitamin E), PIVKA-II | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Sagel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- The Children's Hospital, Aurora, Colorado, United States

REFERENCES:
- [Result] Sagel SD, Sontag MK, Anthony MM, Emmett P, Papas KA. Effect of an antioxidant-rich multivitamin supplement in cystic fibrosis. J Cyst Fibros. 2011 Jan;10(1):31-6. doi: 10.1016/j.jcf.2010.09.005. Epub 2010 Oct 20. PMID 20961818